CLINICAL TRIAL: NCT03535961
Title: Phase II Single Arm Study of Apatinib Combined With Oral Etoposide in Metastatic HER2 Negative Breast Cancer
Brief Title: Apatinib Combined With Oral Etoposide in Metastatic HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-055
Record Dates: First submitted 2017-09-10; First posted 2018-05-24 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib+oral etoposide (Other): apatinib 425/500mg qd, 21days/cycle oral etoposide 50mgmg/m2 d1-10 21days/cycle
  Interventions: Drug: apatinib+oral etoposide

INTERVENTIONS:
Drug: apatinib+oral etoposide — apatinib 425/500mg qd, 21days/cycle oral etoposide 50mgmg/m2 d1-10 21days/cycle

SUMMARY:
The hypothesis of this study is to discover if the all-oral therapy with apatinib plus oral Etoposide can shrink or slow the growth of pretreated HER2 negative metastatic breast cancer.

DETAILED DESCRIPTION:
Apatinib is an orally administered second-generation blocker of the phosphorylation of the tyrosine residues within the intracellular domain of VEGF receptor 2 (VEGFR2). A prospective, open label, phase II multicenter trial of apatinib in heavily pretreated patients with metastatic triple-negative breast cancer demonstrated that the daily dose of apatinib 500 mg/day is active in pretreated metastatic TNBC with encouraging rates of disease stabilization and PFS.

Etoposide is a highly active drug in the treatment of MBC, both as a single agent or in combination regimens, and is well tolerated, with a low incidence of severe toxicity. Clinical trials demonstrated oral Etoposide provided comparable effectiveness to iv Etoposide. and oral availability allows using different schedules.

The NCCN guideline introduces that combination chemotherapy is one of the standard treatment options in metastatic breast cancer, especially in patients with visceral metastases and/or need of rapid symptom or disease control.

Theoretically, anti-angiogenesis regimen combined with chemotherapy may present increasing therapeutic effect. Related researches are urgently needed to find optimal combined therapy.

The hypothesis of this study is to discover if the all-oral therapy with apatinib plus oral Etoposide can shrink or slow the growth of pretreated HER2 negative breast cancer. The safety of the combination will also be studied. Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if this combination is safe and effective in pretreated HER2 negative metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 year-old women; HER2 negative(immunohistochemistry or fluorescence in situ hybridization);
* ECOG score: 0-1, expected survival time ≥ 3months;
* Pathologically or cytologically confirmed breast cancer;
* Anthracycline- / taxane- pretreated (adjuvant, neoadjuvant) breast cancer patients who have failed from 1-2 standard chemotherapies after recurrence and metastasis;
* According to RECIST 1.1, exist at least ≥1 measurable lesion(CT >1cm，other examination >2cm);
* The patients have enough organ function. The laboratory test indexes must comply with the following requirements:

  * Blood routine: neutrophil≥1.5G/L, platelet count ≥80G/L, hemoglobin ≥90g/L
  * Liver function: serum bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤2.5 times the upper limit of normal value; ALT and AST≤5 times the upper limit of normal value when liver metastasis
  * Renal function: serum creatinine ≤ 1.0times the upper limit of normal value, creatinine clearance >50ml/min（Cockcroft-Gault formula)
* Women of child-bearing age should be carried out pregnancy test (serum or urine) within 7 days before recruit, the results should be negative; and are willing to adopt the appropriate methods of contraception during the trial and 8 weeks after last administration；
* Can swallow oral drugs;
* The patients have good compliance to the therapy and follow-up to be scheduled and are able to understand the study protocol and sign the Informed Consent Form.

Exclusion Criteria:

* The patients in pregnancy or lactation growth period and did not take effective contraception;
* The patients who received ≥3 chemotherapies（Do not include endocrine therapy）after recurrence and metastasis; involved in other clinical trials four weeks prior to the start of the study;
* The patients with a variety of factors that affect the oral administration and absorption of drugs;
* The patients previously received anti-VEFG of anti-VEGFR therapies;
* The patients with rapid progression of viscera invasion(liver lesion >1/2 viscera area or liver dysfunction);
* The patients have uncontrollable mental illness.
* The patients who had serious adverse effect to oral etoposide or were allergic to etoposide.
* The patients who have only bone metastasis without other measurable lesion;
* The patients experience severe cardiovascular diseases;
* The patients experience severe upper gastrointestinal ulcer or malabsorption syndrome.
* Abnormal bone marrow functions(neutrophil<1.5G/L, platelet count <75G/L, hemoglobin <90g/L);
* Abnormal renal function(serum creatinine > 1.5 times the upper limit of normal value);
* Abnormal liver function(serum bilirubin ≤ 1.5 times the upper limit of normal value);
* The patients have uncontrollable brain metastasis;
* The patients do have good compliance to the therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
objective response rate(ORR) | up to 1 year after the last patient enrolled
  Objective response rate defined as confirmed complete response or partial response under RECIST 1.1 criteria. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met.

SECONDARY OUTCOMES:
disease control rate(DCR) | through study completion, an average of 1 year
  Number of participants with stable disease or partial response or complete response treating by anloitnib according to RESIST criteria v1.1.
Progression free survival (PFS) | From date of enrollment until the date of first documented progression, assessed up to 24 months
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
overall survival(OS) | From date of enrollment until death, assessed up to 24 months
  OS, defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 1 year
  All the treatment-related adverse events occurred as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Hu N, Zhu A, Si Y, Yue J, Wang X, Wang J, Ma F, Xu B, Yuan P. A Phase II, Single-Arm Study of Apatinib and Oral Etoposide in Heavily Pre-Treated Metastatic Breast Cancer. Front Oncol. 2021 Feb 15;10:565384. doi: 10.3389/fonc.2020.565384. eCollection 2020. PMID 33659204